CLINICAL TRIAL: NCT00918138
Title: A 4-Week, Multicenter, Randomized, Double-Blind, Phase 3b Trial to Evaluate the Efficacy of Saxagliptin in Combination With Metformin XR 1500 mg Versus Up-titrated Metformin XR to 2000 mg in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet and Exercise and a Stable Dose of Metformin XR 1500 mg
Brief Title: Study To Evaluate 24 Hour Blood Sugar Control (24-hour Mean Weighted Glucose) In Subjects That Are Taking Saxagliptin 5 mg Added Onto Metformin XR 1500 XR mg Compared To Subjects Taking Metformin XR 1500 mg Up-titrated To Metformin XR 2000 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV181-085
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2011-10-06 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin + Metformin XR + matching Metformin XR placebo (Experimental): (Saxagliptin 5 mg plus Metformin XR 1500 plus matching Metformin XR 500 mg placebo)
  Interventions: Drug: Saxagliptin; Drug: Metformin XR; Drug: Placebo matching Metformin XR
- Metformin XR + Metformin XR + matching Saxagliptin placebo (Active Comparator): (Metformin XR 500 mg plus Metformin XR 1500 mg plus matching Saxagliptin 5 mg placebo)
  Interventions: Drug: Metformin XR; Drug: Placebo matching Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — Tablets, Oral, 5 mg, once daily, 4 weeks
  Other Names: BMS-477118; Onglyza
  Arms: Saxagliptin + Metformin XR + matching Metformin XR placebo
Drug: Metformin XR — Tablets, Oral, 1500 mg, once daily, 4 weeks
  Other Names: Glucophage XR®
Drug: Placebo matching Metformin XR — Tablets, Oral, 0 mg, once daily, 4 weeks
  Arms: Saxagliptin + Metformin XR + matching Metformin XR placebo
Drug: Metformin XR — Tablets, Oral, 500 mg, once daily, 4 weeks
  Other Names: Glucophage XR®
  Arms: Metformin XR + Metformin XR + matching Saxagliptin placebo
Drug: Placebo matching Saxagliptin — Tablets, Oral, 0 mg, once daily, 4 weeks
  Arms: Metformin XR + Metformin XR + matching Saxagliptin placebo

SUMMARY:
The purpose of this study was to compare effect of Saxagliptin as add-on to Metformin on 24-hour mean weighted glucose (MWG) to the effect of uptitrating Metformin in subjects with T2DM inadequately controlled on metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* 18-78 years of age
* Taking stable dose of metformin immediate release (IR) or XR ≥850 mg and ≤1500 mg as monotherapy for at least 8 weeks prior to screening
* Glycosylated hemoglobin A1C (A1C) 7.5-11.5% at screening
* Fasting C-peptide: ≥1.0 ng/mL
* FPG≥126 mg/dl obtained at the Day -7 visit
* Body mass index (BMI): ≤ 40kg/m²
* A1C ≥ 7.0% and ≤ 11.0% obtained at the Day -7 visit for randomization

Exclusion Criteria:

* Women of childbearing potential unable or unwilling to use acceptable birth control
* Women who are pregnant or breastfeeding
* Significant cardiovascular history
* Active liver disease
* Renal impairment

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (12):
  - Dedicated Phase I, Inc., Phoenix, Arizona
  - Pacific Sleep Medicine Services (Avastra Clinical Trials), Redlands, California
  - Orange County Research Center, Tustin, California
  - Clinical Research Of South Florida, Coral Gables, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - River Birch Research Alliance, Llc, Blue Ridge, Georgia
  - Jasper Clinic, Inc., Kalamazoo, Michigan
  - Clinilabs, Inc., New York, New York
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - Clinical Trials Of Texas Inc., San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
- Israel (4):
  - Local Institution, Beersheba
  - Local Institution, Holon
  - Local Institution, Kfar Saba
  - Local Institution, Safed
- Mexico (2):
  - Local Institution, Durango, Durango
  - Local Institution, Monterrey, Nuevo León

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 219 participants were enrolled; 126 entered single-blind dietary/exercise/metformin extended release (XR) lead-in period (either 4- or 8-weeks long, based on pre-enrollment metformin dose). 33 participants did not enter treatment period (22 no longer met study criteria, 7 withdrew consent, 2 lost to follow-up, 1 adverse event, and 1 other reason).
Groups:
- Saxagliptin 5 mg + Metformin XR 1500 mg: saxagliptin 5 mg plus metformin XR 1500 plus matching metformin XR 500 mg placebo
- Metformin 2000 mg: metformin XR 500 mg plus metformin XR 1500 mg plus matching saxagliptin 5 mg placebo
Period: Overall Study
Arm/Group | Saxagliptin 5 mg + Metformin XR 1500 mg | Metformin 2000 mg
Started | 46 | 47
Completed | 44 | 46
Not Completed | 2 | 1
Not completed — Subject withdrew consent | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 5 mg + Metformin XR 1500 mg | Metformin 2000 mg | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.89 (9.41) | 50.64 (9.74) | 52.25 (9.66)
Age, Customized [Number; unit: participants]
  <65 years | 40 | 45 | 85
  >=65 years | 6 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 21 | 25 | 46
Race/Ethnicity, Customized [Number; unit: Participant]
  White | 43 | 45 | 88
  Black/African American | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: Participant]
  Hispanic/Latino | 16 | 17 | 33
  Not Hispanic/ Not Latino | 8 | 8 | 16
  Not Reported | 22 | 22 | 44
Age categorization Females Only [Number; unit: participants]
  <= 50 years | 5 | 9 | 14
  > 50 years | 16 | 16 | 32
Weight [Mean (Standard Deviation); unit: kg] | 91.27 (18.43) | 86.94 (15.24) | 89.09 (16.94)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.45 (5.08) | 31.06 (4.28) | 31.75 (4.72)
BMI Categorization [Number; unit: Participants]
  < 30 kg/m^2 | 16 | 17 | 33
  >= 30 kg/m^2 | 30 | 30 | 60
Glycosylated Hemoglobin (A1C) [Mean (Standard Deviation); unit: percentage] | 8.6 (0.9) | 8.4 (0.9) | 8.5 (0.9)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — The fasting value is collected at time -30 minutes prior to morning meal
  mg/dL | 163.5 (32.32) | 164.2 (36.21) | 163.8 (34.16)
FPG Categorization [Number; unit: participants] — The fasting value is collected at time -30 minutes prior to morning meal
  participants
    < 126 mg/dL | 5 | 5 | 10
    >= 126 mg/dL to < 150 mg/dL | 11 | 14 | 25
    >= 150 mg/dL to < 220 mg/dL | 28 | 23 | 51
    >= 220 mg/dL to < 300 mg/dL | 2 | 5 | 7
120-minute postprandial glucose (PPG) [Mean (Standard Deviation); unit: mg/dL] — The 120-minute value is collected 120 minutes after start of evening meal
  mg/dL | 281.3 (51.59) | 283.3 (66.14) | 282.3 (59.08)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-Hour Mean Weighted Glucose (MWG) at Week 4
Description: Adjusted mean change from baseline in MWG achieved with saxagliptin 5 mg plus metformin XR versus placebo plus metformin XR at Week 24. MWG was calculated as the area under the curve (AUC) for the full 24 hours expressed as average mg/dL. Glucose measurements were collected 30 minutes before and just prior to each meal (0 minutes) and 30, 60, 120, and 180 minutes after each meal (with 1 additional measurement at 240 minutes after the evening meal), midnight, 3 AM, and at end-of-domicile visit 24 hours after the first measurement. Mean change from baseline was adjusted for baseline value.
Time Frame: Baseline, Week 4
Population: Randomized participants who had both baseline and Week 4 assessments.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin XR 1500 mg | Metformin 2000 mg
Number analyzed (Participants) | 43 | 44
mg/dL
  Baseline Mean | 191.3 (6.26) | 192.0 (6.14)
  Week 4 Mean | 173.2 (5.85) | 184.2 (6.52)
  Adjusted Change from Baseline | -19.0 (5.69) | -8.2 (5.96)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin XR 1500 mg vs Metformin 2000 mg; With at least 36 participants per treatment group (72 total), there is 90% power to detect a difference of 18 mg/dL between the two treatment groups. Assuming approximately 20% of participants will discontinue without any valid post-randomization assessment at Week 4, a total of 90 participants (45 participants per treatment group) needed to be randomized; Test type: Superiority or Other; p = 0.1278, ANCOVA — Comparison between saxagliptin 5 mg + metformin 1500 mg and metformin 2000 mg significant at alpha =0.05 according to sequential testing procedure; Change from baseline to week 4 was analyzed with ANCOVA including treatment group, baseline value and country in the model; Mean Difference (Final Values) = -10.8, 95% CI 2-sided [-24.8 to 3.2], Standard Error of Mean 7.01 — Estimate = adjusted mean change for saxagliptin 5 mg + metformin 1500 mg - adjusted mean change for metformin 2000 mg

2. Secondary Outcome: Change From Baseline to Week 4 in 2-hour Postprandial Glucose (PPG) (2 Hours After the Evening Meal)
Description: Adjusted mean change from baseline in 2-hour postprandial (after mealtime) plasma glucose two hours after start of the evening meal during 24-hour domicile visits evaluated both at pre-randomization (baseline) and at Week 4. Mean change from baseline was adjusted for baseline value.
Time Frame: Baseline, Week 4
Population: Randomized participants who had both baseline and Week 4 assessments.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin XR 1500 mg | Metformin 2000 mg
Number analyzed (Participants) | 44 | 46
mg/dL
  Baseline mean | 229.7 (9.07) | 234.0 (10.32)
  Week 4 mean | 195.3 (7.99) | 228.1 (11.30)
  Adjusted mean change from baseline | -31.4 (9.69) | -0.2 (10.09)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin XR 1500 mg vs Metformin 2000 mg; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -31.1, 95% CI 2-sided [-54.6 to -7.7], Standard Error of Mean 11.80 — Estimate = adjusted mean change for saxagliptin 5 mg + metformin 1500 mg - adjusted mean change for metformin 2000 mg

3. Secondary Outcome: Change From Baseline Fasting Plasma Glucose (FPG) at Week 4, Obtained Immediately Before the Morning Meal
Description: FPG measurements were done at baseline, day 14 and 28. At baseline and day 28, the FPG value=plasma glucose value collected 30 minutes prior to the morning meal during the domicile visit.
Time Frame: Baseline, Week 4
Population: Randomized participants who had both baseline and Week 4 assessments. Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin XR 1500 mg | Metformin 2000 mg
Number analyzed (Participants) | 45 | 47
mg/dL
  Baseline mean | 162.9 (4.84) | 164.2 (5.28)
  Week 4 LOCF mean | 155.2 (6.49) | 161.8 (5.23)
  Adjusted mean change from baseline | -9.3 (5.93) | -3.6 (6.17)
Statistical Analysis 1: Comparison: Saxagliptin 5 mg + Metformin XR 1500 mg vs Metformin 2000 mg; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-20.0 to 8.5], Standard Error of Mean 7.18 — Estimate = adjusted mean change for saxagliptin 5 mg + metformin 1500 mg - adjusted mean change for metformin 2000 mg

4. Other Pre Specified Outcome: Participants With Confirmed Hypoglycemia Events During the Treatment Period
Description: 'Confirmed' = recorded on the hypoglycemia AE case report form with a fingerstick for glucose <= 50 mg/dL and associated symptoms.
Time Frame: AEs: up to last treatment day (LTD) +1 day or last visit day (LVD), whichever came last ; SAEs: up to LTD +30 days or LVD + 30 days, whichever came last. Mean duration of exposure=27.7 days for Saxa 5 mg + Met XR 1500 mg, and 28.3 days for Met 2000 mg.
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Saxagliptin 5 mg + Metformin XR 1500 mg | Metformin 2000 mg
Number analyzed (Participants) | 46 | 47
participants | 0 | 0

5. Other Pre Specified Outcome: Participants With Reported Hypoglycemic Adverse Events During Treatment Period
Description: Hypoglycemic events are based upon the Saxagliptin Predefined List of Events, which includes hypoglycemia, blood glucose decreased, and hypoglycemic unconsciousness. The Hypoglycemic events occurred in less than 5% of the participants and hence do not appear in the adverse events module.
Time Frame: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Saxagliptin 5 mg + Metformin XR 1500 mg | Metformin 2000 mg
Number analyzed (Participants) | 46 | 47
participants | 1 | 2

ADVERSE EVENTS:
Arm/Group | Metformin 2000 mg | Saxagliptin 5 mg + Metformin XR 1500 mg
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/46
Other Adverse Events (participants affected / at risk) | 0/47 | 3/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin 2000 mg (N=47) | Saxagliptin 5 mg + Metformin XR 1500 mg (N=46)
DEATH (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin 2000 mg (N=47) | Saxagliptin 5 mg + Metformin XR 1500 mg (N=46)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.